CLINICAL TRIAL: NCT03238469
Title: Long-term Efficacy and Safety of Microwave Ablation in the Treatment of Mild Axillary Hidradenitis Suppurativa
Brief Title: Microwave Ablation in Mild Axillary Hidradenitis Suppurativa
Acronym: WAVE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Negative clinical outcomes
Sponsor: M.B.A. van Doorn (Other)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Sponsor-Investigator, M.B.A. van Doorn, MD, PhD, Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WAVE trial
Record Dates: First submitted 2017-07-31; First posted 2017-08-03 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Hidradenitis Suppurativa; Acne Inversa
Keywords: Microwave Ablation; Hair Follicle; Sweat gland
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Intervention Model Description: Randomized intra-patient controlled trial.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Microwave ablation (Experimental): One-sided single microwave ablation (MWA) treatment in one axillary region with a miraDry device.
  Interventions: Device: Microwave ablation
- No microwave ablation (No Intervention): Lesion intervention in the non-MWA treated contralateral axilla consists of once daily topical clindamycin 1% lotion.

INTERVENTIONS:
Device: Microwave ablation — A one-sided (either right or left axillary area) single MWA treatment using a miraDry system. The miraDry device has a microwave output frequency of 5.8 GHz and microwave energy level settings ranging from 1 to 5, corresponding with a delivery time in seconds between 2.40 sec and 3.00 sec. For this study standard 5 (i.e. 3.00 sec) is set as treatment setting.
  Arms: Microwave ablation

SUMMARY:
With microwave ablation (MWA), using the heat generated from electromagnetic waves in the microwave energy spectrum, hair follicles and apocrine glands in the (hypo)dermis are ablated through thermolysis. MWA was recently approved for the treatment of axillary hyperhidrosis (miraDry) and removal of axillary hair (miraSmooth). By permanent removal of hairs and sweat glands, the investigators hypothesize a beneficial and long-term sustainable preventive effect of MWA in HS patients.

DETAILED DESCRIPTION:
Hidradenitis suppurativa (HS) is a chronic, inflammatory skin disease of the hair follicle, and is predominantly located in the axillary, inguinal and anogenital regions. Current treatment options for HS include systemic oral antibiotics, anti-TNFα, and surgery, which are used to treat the consequences rather than treating the primary pathogenesis of HS. With microwave ablation (MWA), using the heat generated from electromagnetic waves in the microwave energy spectrum, hair follicles, eccrine and apocrine glands in the (hypo)dermis are ablated through thermolysis. MWA was recently approved for the treatment of axillary hyperhidrosis (miraDry) and removal of axillary hair (miraSmooth). By permanent removal of hairs and sweat glands, the investigators hypothesize a beneficial and long-term sustainable preventive effect of MWA in HS patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years of age) male or female patients with mild HS and able to participate, willing to give written informed consent and to comply with the study restrictions;
* Minimum of 3 AN-count located in each axilla;
* Maximum of 5 AN-count located in each axilla.

Exclusion Criteria:

* Patients with >1 abscesses or draining fistulas per axillary region;
* AN-count ≥ 5 in other regions than the axillary area;
* Any current and / or recurrent clinically significant skin condition in the treatment area other than HS;
* Surgical scars covering more than 25% of each individual axillary area;
* Open surgical wound(s) in the axillary areas prior to randomization;
* Use of anti-inflammatory or immunomodulatory medication (intralesional corticosteroids, oral antibiotics, biologics, prednisone) within 2 weeks prior to randomization;
* Contraindication for miraDry therapy;
* Heart pacemakers and other electronic device implants;
* Supplemental oxygen;
* Resistance to or history of intolerance of local anesthesia including lidocaine and epinephrine;
* Previous use of miraDry therapy or MWA in the axillary area;
* Previous use of successful laser or light therapy for hair removal in the axillary area;
* Use of botulinum toxin injections 6 months prior to randomization;
* Use of aluminiumhydroxychloride 1 month prior to randomization;
* Pregnant or lactating women at randomization.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Hidradenitis Suppurativa Clinical Response (HiSCR50) | 6 months
  The proposed definition of 50% responders to treatment (HiSCR50 achievers) is: (i) at least a 50% reduction in ANs, (ii) no increase in the number of abscesses, and (iii) no increase in the number of draining fistulas from baseline

SECONDARY OUTCOMES:
Hidradenitis Suppurativa Clinical Response (HiSCR30) | 6 months
  The proposed definition of 30% responders to treatment (HiSCR30 achievers) is: (i) at least a 30% reduction in ANs, (ii) no increase in the number of abscesses, and (iii) no increase in the number of draining fistulas from baseline
Patient-reported number of HS flares | 6 months
  The number of HS flares in the treated and untreated axillae. At baseline retrospective assessment on last month, and during follow-up prospective assessment using a diary where patients will report the number of acute boils per axilla.
Average number of hair containing follicles | 6 months
  Dermatoscopy of three fields per axilla
Extent of sweat production | 6 months
  Starch-Iodine test per axillary region
Patient-reported pain and pruritus | 6 months
  Numerical rating scale (NRS) to assess pain and itch per axillary region
Incidence of (treatment-emergent) adverse events | 6 months
  Safety and tolerability of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Errol Prens, MD, PhD, Principal Investigator — Professor
Locations (1):
- Erasmus University Medical Center, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No
metc@erasmusmc.nl